CLINICAL TRIAL: NCT03735212
Title: A Regional Partnership for New York City to Improve Child Welfare Outcomes Among Pregnant Women at Risk of Substance Misuse and Their Newborns
Brief Title: Regional Partnership for Pregnant Women at Risk of Substance Misuse and Their Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-9611; 90CU-0102-01-00 (Other Grant/Funding Number: New York Children's Bureau)
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program Group (Experimental): Participants in this group receive enhanced services as the intervention. These services include Motivational Enhancement, Incredible Years, and Contingency Management. Participants also receive case management services to support referrals to substance use.
  Interventions: Behavioral: Enhanced Services
- Control Group (No Intervention): Participants in this group receive services as usual.

INTERVENTIONS:
Behavioral: Enhanced Services — Participants receive enhanced services over a period of 6 months to support substance abuse recovery, referral to treatment, and parenting skills.
  Arms: Program Group

SUMMARY:
This study recruits pregnant women and new mothers who are at risk of substance use concerns during pregnancy or delivery. These women are followed for 6 months and randomized into two groups; they may receive services as usual, or enhanced services. Enhanced services include evidence based interventions and case management to support referrals to substance abuse treatment, and to teach strategies specifically targeted to parenting newborns.

DETAILED DESCRIPTION:
The dual goals of this project are to (i) improve communication and collaboration between substance abuse treatment providers, obstetricians, and child welfare providers, and (ii) to enhance child welfare outcomes for pregnant women who are at risk of substance misuse and their babies. There is a particular need for a partnership in this area as New York State implements the 2016 Comprehensive Addiction and Recovery Act (CARA) legislation, which focuses on a multi-agency approach to the problem of substance abuse for families at risk of child welfare involvement.

Services are delivered through Montefiore's Department of Obstetrics & Gynecology and Women's Health (Obstetrics). Mothers-to-be who have screened at risk or tested positive for substances will be randomly assigned to receive services as usual as part of the comparison group, or to receive enhanced prenatal services as part of the program group. Program services include 3 empirically supported interventions: Motivational Enhancement to enhance intrinsic motivation to change unhealthy behaviors and support their referral to substance abuse treatment; Incredible Years to improve parenting skills, especially related to infancy and early childhood; and Contingency Management to reinforce healthy behaviors, including attendance at treatment and abstinence.

Women enrolled into the study are randomly assigned into a program or comparison group. Parent, child, and family outcomes are evaluated using self-report and administrative data.

ELIGIBILITY:
Inclusion Criteria:

-The potential subject: (i) is a woman who receives prenatal care at Montefiore Medical Center, (ii) is at least 16 weeks pregnant and at most 12 weeks post-partum, and (iii) is identified as at-risk for substance use, and/or has tested positive for at least one substance.

Exclusion Criteria:

* Minors
* Those who are less than 16 weeks pregnant or more than 12 weeks post-partum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change in composite Addiction Severity Index (ASI) score from baseline | Change between Baseline and Follow up (6 month interval)
  ASI is an assessment tool which will be administered to participants to evaluate their condition in 7 key problem areas of substance use and addiction severity (i.e, medical status, employment, drug use, alcohol use, legal status, family/social status, psychiatric status). Questions generally have a score of 0 of 1 associated. For example, if the patient answers yes, they may score 1; if they answer no, they may score 0. For some items, the scoring may be reversed.
  0-1: No imminent problem, treatment not indicated. 2-3: Slight problem; treatment may not be necessary. 4-5: Moderate problem, a treatment plan should be considered. 6-7: Considerable difficulty, begin a treatment plan. 8-9: Extreme problem, treatment is vital.
  Composite scores will be used to assign a severity rating. The higher the score, the higher the need for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wetzler, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data with other researchers.